CLINICAL TRIAL: NCT07375524
Title: A Phase 2 Study on the Safety and Efficacy of the Anti-BAFF-R Monoclonal Antibody, ESG206, in Patients With Primary Sjogren Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Escugen Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESG206-PSS-01
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Primary Sjögren Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESG206 Low Dose (Active Comparator): ESG206 Low Dose Injection administered by intravenous infusion
  Interventions: Drug: ESG206
- ESG206 High Dose (Active Comparator): ESG206 High Dose Injection administered by intravenous infusion
  Interventions: Drug: ESG206
- Placebo (Placebo Comparator): Placebo Injection administered by intravenous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ESG206 — ESG206 Low Dose administered by intravenous infusion
  Arms: ESG206 High Dose
Drug: ESG206 — ESG206 High Dose administered by intravenous infusion
  Arms: ESG206 Low Dose
Drug: Placebo — Placebo administered by intravenous infusion
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase II study designed to evaluate the efficacy and safety of ESG206 in participants with primary Sjögren's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age) with a confirmed diagnosis of primary Sjögren's syndrome according to the 2016 American College of Rheumatology (ACR) / European League Against Rheumatism (EULAR) classification criteria.
* Evidence of active disease at screening
* Willing and able to provide written informed consent

Exclusion Criteria:

* Secondary Sjögren's syndrome or other clinically significant autoimmune or inflammatory diseases
* Prior or recent use of prohibited immunomodulatory therapies
* Clinically significant infections, malignancies, or uncontrolled medical conditions
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in ESSDAI score compared with placebo. | Up to approximately 25 weeks
  ESSDAI is a validated clinical disease activity index for Sjögren's syndrome. It includes 12 organ-specific domains, each scored by the investigator according to severity using 3- or 4-level scales. Weighted domain scores are summed to generate a total score (maximum score: 123). Domains include constitutional, lymphadenopathy, glandular, articular, cutaneous, pulmonary, renal, muscular, peripheral nervous system, central nervous system, hematological, and biological domains. Higher scores on the ESSDAI scale are associated with poorer health states.

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - Changde First People's Hospital, Changde, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - the Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Huzhou Third People's Hospital, Huzhou, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Wenzhou People's Hospital, Wenzhou, Zhejiang